CLINICAL TRIAL: NCT03065010
Title: A Multicenter Open-label Non-comparative 2-Stage Phase 1a/1b Study to Assess the Safety and Pharmacokinetics of BCD-115 (JSC BIOCAD, Russia) in Combination With Endocrine Therapy in Women With ER(+) HER2(-) Local Advanced and Metastatic Breast Cancer
Brief Title: Study of BCD-115 in Women With ER(+) HER2(-) Local Advanced and Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-115-1
Record Dates: First submitted 2017-02-16; First posted 2017-02-27 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD-115 in dose escalation regimen (Other): BCD-115 will be administered p.o. with intrapatient dose escalation in the population of patients with ER(+) HER2(-) advanced breast cancer in combination with a standard dose of endocrine therapy.
  Interventions: Drug: BCD-115

INTERVENTIONS:
Drug: BCD-115 — Inhibitor of CDK8/19

SUMMARY:
A Multicenter Open-label Non-comparative 2-Stage Phase 1a/1b Study to Assess the Safety and Pharmacokinetics of Oral BCD-115 (JSC BIOCAD, Russia) in Combination with Endocrine Therapy in Women with ER(+) HER2(-) Local Advanced and Metastatic Breast Cancer

DETAILED DESCRIPTION:
Multicentre dose-finding open-label non-comparative phase Ia/Ib clinical trial for investigation of the safety, tolerability, pharmacokinetics of BCD-115 administered p.o. with intrapatient dose escalation in the population of patients with ER(+) HER2(-) advanced breast cancer in combination with a standard dose of endocrine therapy.

The trial will be conducted in two stages:

Stage 1 - finding of the maximum tolerated dose, determination of the recommended dose for Stage 2.

Stage 2 - study of the recommended dose from Stage 1 of BCD-115, analysis of tolerability and safety of selected dose/doses in additional cohorts, and determination of the estimated therapeutic dose/doses for further clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and ability to follow the Protocol procedures;
2. Age ≥18 years;
3. Female gender;
4. Postmenopausal status (Prior bilateral surgical oophorectomy; or medically confirmed post-menopausal status defined as spontaneous cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause);
5. Histologically proven diagnosis of adenocarcinoma of the breast with evidence of metastatic disease;
6. Progression of advanced breast cancer on first line endocrine therapy for advanced breast cancer.
7. ER positive tumor ≥ 10%;
8. HER2 negative breast cancer by FISH or IHC;
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
10. Measurable disease according to RECIST 1.1 (only bone disease is not allowed)
11. Resolution of all acute toxic effects of prior therapy (including endocrine therapy) or surgical procedures to CTCAE grade ≤1
12. Adequate organ function;
13. Life expectancy - 12 weeks or more from the moment of randomization

Exclusion Criteria:

1. HER2-positive tumour ;
2. Patients with unstable brain metastases, advanced, symptomatic, visceral spread disease, that are at risk of life-threatening complications in the short term (including patients with massive uncontrolled effusions pleural, pericardial, peritoneal, pulmonary lymphangitis, and over 50% liver involvement).
3. Important cardiovascular events in the past 6 months to randomization;
4. GI diseases which may affect the absorption of the study drug;
5. Inadequate hematopoietic function: neutrophils ≤1500/mm3, platelets ≤100 000/mm3,or hemoglobin ≤90 g/L;
6. Inadequate renal function: creatinine level ≥ 1.5 × upper limit of normal (ULN);
7. Inadequate liver function: bilirubin level ≥ 1.5 × ULN, AST and ALT levels ≥ 2.5 × ULN (5 × ULN for patients with liver metastases), alkaline phosphatase level ≥ 5 × ULN;
8. Concurrent antitumor treatment 21 days before randomization (surgery, radiation therapy; chemotherapy, except endocrine therapy);
9. Any other concomitant cancer including contralateral breast cancer revealed within 5 years prior to screening, except curatively treated intraductal carcinoma in situ, curatively treated cervical carcinoma in situ or curatively treated basal cell or squamous cell carcinoma;
10. Conditions limiting patient's adherence to protocol requirements (dementia, neurologic or psychiatric disorders, drug addiction, alcoholism and others);
11. Concomitant participation in other clinical trials, previous participation in other clinical trials within 30 days before entering into the trial, previous participation in the same trial;
12. Acute or active chronic infections;
13. HCV, HBV, HIV or syphilis infections;
14. Obstacles to p.o. administration of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Femaile gender
Enrollment: 6 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC0-t) | 90 days
  To determine AUC0-t after single doses of BCD-115 p.o. administration with dose escalation;
Peak Plasma Concentration (Cmax) | 90 days
  To determine observed maximum concentration in plasma or serums after single doses of BCD-115 p.o. administration with dose
The incidence and severity of AEs | 90 days
  The incidence and severity of AEs (%) related with the therapy based on results of review by 3 experts (%)
The incidence of grade 3-4 AEs | 90 days
  The incidence of grade 3-4 AEs (%) related with the therapy based on results of review by 3 experts

SECONDARY OUTCOMES:
Treatment discontinuation due to adverse events | 90 days
  Treatment discontinuation due to adverse events (%)

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin Russian Cancer Research Center, Saint Petersburg, Russia